CLINICAL TRIAL: NCT04239768
Title: Efficacy and Tolerance Evaluation of an Antiage Aesthetic Treatment for the Middle and Inferior Third of the Face
Brief Title: Efficacy of an Antiage Aesthetic Treatment for the Middle and Inferior Third of the Face
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Derming SRL (Other)
Responsible Party: Principal Investigator, Adele Sparavigna, Principal Investigator, Derming SRL
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E0919
Record Dates: First submitted 2020-01-21; First posted 2020-01-27 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Face Skin Laxity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MonoDermà HA gel combined to a low level laser (Experimental): "Monodermà HA Bio-revitalizing gel" is a sterile, biodegradable, isotonic intradermal filler produced by Innate S.r.l. (Italy) and distributed by Giuliani S.p.A. (Italy) in non-pyrogenic pre-filled syringe of 2 ml containing 2% (20mg/ml) of medium chain (1.0-1.5 x 106 Dalton) hyaluronic acid (HA), obtained from bacterial fermentation, in a physiologic buffer (see Appendix 1) and used as a filler for the correction of deep skin sagging and roughness.
  Interventions: Device: MonoDermà HA gel combined to a low level laser

INTERVENTIONS:
Device: MonoDermà HA gel combined to a low level laser — Two intradermal injections of the filler were performed during the basal and after 1 month, on the middle and inferior third of the face (1ml for each face side) using a needle (30G).
  Immediately after both injection procedures, LLLT session were performed on the same face area for a total of 8 minutes, using three different wavelengths (450 nm, 650 nm and 1064 nm) simultaneously.

SUMMARY:
Primary endpoint of the study is to evaluate clinically and by non-invasive instrumental evaluations the aesthetic performance, on the third middle and inferior of the face, of "MonoDermà HA Bio-revitalizing gel", an intradermal filler containing hyaluronic acid, combined to a low level laser therapy (LLLT) to obtain a stable photo-cross-linking effect inside the dermis.

ELIGIBILITY:
Inclusion Criteria:

* female sex;
* Caucasian race;
* non smokers;
* no alcohol abuse and/or drug use;
* 40-65 years;
* FVLS 2-4 ;
* available and able to return to the study site for the post-procedural follow-up examinations;
* accepting not to change their habits regarding food, physical activity, cosmetic and cleansing products for the face;
* accepting not to expose their face to strong UV irradiation (UV session and/or sun bathes) during the entire duration of the study, without appropriate sun protection;
* accepting to sign the informed consent form.

Exclusion Criteria:

* Pregnancy (only for female subjects not in menopause);
* lactation (only for female subjects not in menopause);
* smokers;
* alcohol abuse and/or drug use;
* female subjects not in menopause, who do not use adequate contraceptive precautions in order to avoid pregnancies during the study;
* female subjects not in menopause, who do not accept to perform the pregnancy test at T0 and T1 (before the 1st and the 2nd aesthetic procedure);
* Body Mass Index (BMI) variation (± 1) during the study period;
* having performed face treatments for aesthetic correction (biomaterials implants, face lifting, botox injections, laser, chemical peeling) in the 6 months beginning of the study;
* having used permanent filler in the past;
* change in the normal habits regarding food, physical activity, face cosmetic, cleansing and make-up use during the month preceding the test;
* sensitivity to the test filler or its ingredients, including delayed hypersensitivity to hyaluronic acid and granulomatous reactions (to be assessed by the investigator during the baseline);
* subjects whose insufficient adhesion to the study protocol is foreseeable;
* participation in a similar study currently or during the previous 9 months;
* dermatitis;
* presence of cutaneous disease on the tested area, as lesions, scars, malformations;
* subjects that tend to develop hypertrophic scars;
* recurrent facial/labial herpes;
* clinical and significant skin condition on the test area (e.g. active eczema, psoriasis, severe rosacea, scleroderma, local infections and severe acne);
* diabetes;
* endocrine disease;
* hepatic disorder;
* renal disorder;
* cardiac disorder;
* pulmonary disease;
* cancer;
* neurological or psychological disease;
* inflammatory/immunosuppressive disease;
* drug allergy;
* anticoagulants and antiplatelet drugs, anti-histaminic, topic and systemic corticosteroids, narcotic, antidepressant, immunosuppressive drugs (with the except of contraceptive or hormonal treatment started more than 1 year ago);
* using of drugs able to influence the test results in the investigator's opinion.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2020-01-17 (Actual)

PRIMARY OUTCOMES:
Wrinkle Severity Rating Scale (WSRS) grade variation | Baseline (T0), 1 month (T1), 2 months (T2), 3 months (T3)
  Reduction of wrinkles severity corresponding to a decrease from the baseline of the Wrinkle Severity Rating Scale (WSRS) clinical score where:
  Grade 1 (absent): no visible nasolabial fold; continuous skin line. Grade 2 (mild): shallow but visible nasolabial fold with a slight indentation; minor facial feature.
  Grade 3 (moderate): moderately deep nasolabial folds; clear facial feature visible at normal appearance but not when stretched.
  Grade 4 (severe): very long and deep nasolabial folds; prominent facial feature; <2mm visible fold when stretched.
  Grade 5 (very severe): extremely deep and long nasolabial fold, detrimental to facial appearance; 2-4 mm visible V-shaped fold when stretched.
Facial Volume Loss Scale (FVLS) grade variation | Baseline (T0), 1 month (T1), 2 months (T2), 3 months (T3)
  Reduction of face volume loss corresponding to a decrease from the baseline of the Facial Volume Loss Scale (FVLS) where:
  Grade 1: Mild flattening or shadowing of one or more facial regions (including the cheek, temple, preauricolar and periorbital areas). No prominent bony landmarks. No visibility of underlying musculature.
  Grade 2: An intermediate point between grade 1 and grade 3. Grade 3: Moderate concavity of one or more facial regions (including the cheek, temple, preauricolar and periorbital areas. Prominence of bony landmarks. May have visibility of underlying musculature.
  Grade 4: An intermediate point between grade 3 and grade 5. Grade 5: Severe indentation of one or more facial regions (including the cheek, temple, preauricolar and periorbital areas). Severe prominence of bony landmarks. Clear visibility of underlying musculature.
Photographic documentation (3D pictures) | Baseline (T0), 1 month (T1), 2 months (T2), 3 months (T3)
  Three-dimensional pictures of the face taken by VECTRA H1 handheld imaging system.
Face volume variation | Baseline (T0), 1 month (T1), 2 months (T2), 3 months (T3)
  Face volume image analysis was carried on the 3D pictures taken by Vectra H1 thanks to Vectra analysis module (VAM) software

CONTACTS AND LOCATIONS:
Locations (1):
- DERMING, Milan, MI, Italy